CLINICAL TRIAL: NCT05339477
Title: The Physical Activity Post Myocardial Infarction SWEDEHEART Prospective Cohort Study (ACTIVITY-SWEDEHEART)
Brief Title: The Physical Activity Post Myocardial Infarction SWEDEHEART Prospective Cohort Study
Acronym: ACTIVITY
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Maria Bäck, Professor, physiotherapist, Sahlgrenska University Hospital
Other Study IDs: 277371
Record Dates: First submitted 2022-04-10; First posted 2022-04-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Myocardial Infarction
Keywords: physical activity; Accelerometer; Registry
MeSH Terms: conditions — Myocardial Infarction; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort group: Diagnosis of a type 1 myocardial infarction registered in SWEDEHEART Age 18-79 years at discharge from hospital
  Interventions: Other: Accelerometer measurement

INTERVENTIONS:
Other: Accelerometer measurement — Study personnel will initiate an accelerometer and inform the patient to wear the accelerometer with an elastic belt on their right hip during waking hours for seven consecutive days. Moreover, patients are instructed to register their wear time in an activity diary in paper form. In addition, patients will register their working hours, if relevant. After seven days, patients send back the accelerometer and diary in a pre-paid envelope. The same procedure is repeated at the second follow-up visit at 1 year.

SUMMARY:
The association between objectively measured physical activity intensities (light, moderate and vigorous), sedentary time and clinical outcomes has not been clarified in patients after a myocardial infarction.

The overall objective of the study is to explore associations between accelerometer measured physical activity and clinical outcomes after a myocardial infarction. Moreover, the association between changes in physical activity and outcomes will be assessed.

DETAILED DESCRIPTION:
It is estimated to include 4000 patients with myocardial infarction during 2 years. Patients will wear the accelerometer for 7 days at follow-up visits (2 months and 1 year) after discharge. The investigators will examine the dose-response relations of several exposure variables from the accelerometer measurements with the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosis of a type 1 myocardial infarction registered in SWEDEHEART
* Age 18-79 years at discharge from hospital
* Attending the first visit in the cardiac rehabilitation (CR) registry SEPHIA (2 months after discharge)

Exclusion Criteria:

* Inability to understand Swedish
* Non-ambulatory
* Any mental condition that may interfere with the possibility for the patient to comply with the study protocol

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myocardial infarction will be recruited at the first (2 months after discharge) cardiac rehabilitation follow-up visit at hospital.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2029-04-26 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular event (MACE) | 1 year after the index cardiac event
  The composite incidence of cardiovascular mortality, non-fatal myocardial infarction, non-fatal ischemic stroke, coronary revascularization, hospitalization for new or worsening heart failure

SECONDARY OUTCOMES:
Cardiovascular mortality | 1 year after the index cardiac event
  Incidence of cardiovascular mortality
Non-fatal myocardial infarction | 1 year after the index cardiac event
  Incidence of non-fatal myocardial infarction
Non-fatal ischemic stroke | 1 year after the index cardiac event
  Incidence of non-fatal ischemic stroke
Coronary revascularization | 1 year after the index cardiac event
  Incidence of coronary revascularization
Heart failure | 1 year after the index cardiac event
  Incidence of hospitalization for new or worsening heart failure
Major adverse cardiovascular event (MACE) | 3 years after the index cardiac event
  The composite incidence of cardiovascular mortality, non-fatal myocardial infarction, non-fatal ischemic stroke, coronary revascularization, hospitalization for new or worsening heart failure
Cardiovascular mortality | 3 years after the index cardiac event
  Incidence of cardiovascular mortality
Non-fatal myocardial infarction | 3 years after the index cardiac event
  Incidence of non-fatal myocardial infarction
Non-fatal ischemic stroke | 3 years after the index cardiac event
  Incidence of non-fatal ischemic stroke
Coronary revascularization | 3 years after the index cardiac event
  Incidence of coronary revascularization
Heart failure | 3 years after the index cardiac event
  Incidence of hospitalization for new or worsening heart failure
All-cause death | 1 year after the index cardiac event
  Incidence of all-cause death
All-cause death | 3 year after the index cardiac event
  Incidence of all-cause death

OTHER OUTCOMES:
Smoking status | 1 year after the index cardiac event
  0=Never smoker, 1=Former smoker > 1 month, 2=Smoker
The Swedish Healthy diet questionnaire | 1 year after the index cardiac event
  Four questions with Likert scale 0-3 points. Higher scores indicate better outcomes
Health-related quality of life (EuroQol- 5 Dimension) | 1 year after the index cardiac event
  EuroQol- 5 Dimension (EQ-5D-3L) The EQ-5D-3L comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. Higher scores indicate better outcomes.
Health-related quality of life (EQ visual analogue scale) | 1 year after the index cardiac event
  EQ visual analogue scale (EQ VAS). The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'.
Triglycerides | 1 year after the index cardiac event
  Plasma levels of triglycerides (mmol/L). Higher values indicate worse outcome.
High-density lipoprotein (HDL) cholesterol | 1 year after the index cardiac event
  Plasma levels of HDL (mmol/L). Higher values indicate better outcome
Low-density lipoprotein (LDL) cholesterol | 1 year after the index cardiac event
  Plasma levels of LDL cholesterol (mmol/L). Higher values indicate worse outcome
Hemoglobin A1c (HbA1c) | 1 year after the index cardiac event
  HbA1c (mmol/L). Measures the amount of blood sugar. Higher values indicate worse outcome
Blood pressure | 1 year after the index cardiac event
  mmHg
Body weight | 1 year after the index cardiac event
  kg
Waist circumference | 1 year after the index cardiac event
  cm

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bäck, PhD, Principal Investigator — Department of physiotherapy, Sahlgrenska University Hospital
Locations (35):
- Sweden (35):
  - Alingsås lasarett, Alingsås
  - NU-sjukvården Dalslands sjukhus, Bäckefors
  - Bollnäs sjukhus, Bollnäs
  - Höglandssjukhuset Eksjö, Eksjö
  - Lasarettet Enköping, Enköping
  - Gävle sjukhus, Gävle
  - Sahlgrenska University Hospital Sahlgrenska, Gothenburg
  - Helsingborgs lasarett, Helsingborg
  - Jönköping Ryhov Hospital, Jönköping
  - Kalix sjukhus, Kalix
  - Länssjukhuset Kalmar, Kalmar
  - Centralsjukhuset Karlstad, Karlstad
  - Kullbergska sjukhuset, Katrineholm
  - Västmanlands sjukhus Köping, Köping
  - Universitetssjukhuset Linköping, Linköping
  - Sunderby sjukhus, Luleå
  - NU-sjukvården Lysekil, Lysekil
  - Skåne Universitetssjukhus Malmö, Malmo
  - Vrinnevisjukhuset, Norrköping
  - Oskarshamns sjukhus, Oskarshamn
  - Västmanlands sjukhus Sala, Sala
  - Sandvikens sjukhus, Sandviken
  - Capio Närsjukhus Simrishamn, Simrishamn
  - Skaraborgs sjukhus Skövde, Skövde
  - Söderhamns sjukhus, Söderhamn
  - Capio St Göran, Stockholm
  - Karolinska University Hospital Solna and Huddinge, Stockholm
  - Södersjukhuset, Stockholm
  - NU-sjukvården Strömstad, Strömstad
  - Norrlands Universitetssjukhus Umeå, Umeå
  - Akademiska sjukhuset, Uppsala
  - Hallands sjukhus Varberg, Varberg
  - Värnamo sjukhus, Värnamo
  - Västerviks sjukhus, Västervik
  - Visby Lasarett, Visby